CLINICAL TRIAL: NCT06350656
Title: Study of Cerebral Compliance in Neurosurgical Intensive Care Units (EC2)
Acronym: EC2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN282022/CHUSTE
Record Dates: First submitted 2023-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cerebrospinal; Disorder
Keywords: Cerebrospinal compliance; Intracranial pressure.; Head injury; Pulse waveform
MeSH Terms: conditions — Central Nervous System Diseases; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical data collection — Post-retrieval from the medical record
Other: Therapeutic data collection — Post-retrieval from the medical record
Other: IntraCranial Pression (ICP) values collection — Post-retrieval of ICP values from the monitor

SUMMARY:
Despite the massive use of intracranial pressure in neuro-resuscitation, there is still no cerebral compliance evaluation index used in current practice to guide therapy.

In treatment guidelines for intracranial hypertension, patients are placed in a prone position at about 30 degrees. Several times a day, during nursing care, patients are flattened, which corresponds to a cerebral compliance test by adding a volume of cerebrospinal fluid to the cranial box.

DETAILED DESCRIPTION:
This study aims to analyse the shape of the different components of the intracranial pressure waves (P1, P2, and P3) when the patient is flattened to determine an index to define the level of cerebral compliance.

ELIGIBILITY:
Inclusion Criteria:

* Continuous intracranial pressure monitoring
* Sedated patient on mechanical ventilation

Exclusion Criteria:

* Craniectomy
* Major hemodynamic failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sedated patient on mechanical ventilation with continuous intracranial pressure monitoring
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Intracranial pressure (mmHg) | Year : 1
  Intracranial pressure is measured before (Raising the head by 30°) and during the flattening (Raising the head by 0°).
  Theses measures are done twice a day.
  The mean of theses values is calculated.

SECONDARY OUTCOMES:
Correlation between ICP (Intra Cranial Pressure) doses and cerebral compliance | Year : 1
  Compare the ICP (Intra Cranial Pressure) dose value with the compliance index during the period before or after the flattening

CONTACTS AND LOCATIONS:
Overall Officials: LAURENT GERGELE, MD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (7):
- France (7):
  - CENTRE HOSPITALIER Charponnay, Chaponnay
  - CENTRE HOSPITALIER UNIVERSITAIRE Grenoble, Grenoble
  - HOPITAL NORD La Tronche, La Tronche
  - APHP, Paris
  - Hopital Lariboisiere - Ahph, Paris
  - CENTRE HOSPITALIER UNIVERSITAIRE Rennes, Rennes
  - CENTRE HOSPITALIER UNIVERSITAIRE Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No